CLINICAL TRIAL: NCT01070550
Title: Prospective Observational Study on Predictors of Early On-treatment Response and Sustained Virological Response in a Cohort of Treatment naïve HCV-infected Patients Treated With Pegylated Interferons.
Brief Title: PROPHESYS 1: An Observational Study on Predictors of Response in Treatment-naïve Patients With Chronic Hepatitis C Virus (HCV)Treated With Pegasys (Peginterferon Alfa-2a)
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MV21012
Record Dates: First submitted 2010-02-09; First posted 2010-02-18 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort: Participants chronically infected with the hepatitis C virus including Genotypes 1 to 6.
  Interventions: Drug: Peginterferon alfa-2a (Pegasys®)

INTERVENTIONS:
Drug: Peginterferon alfa-2a (Pegasys®) — Peginterferon (PEG-IFN) alfa-2a Peginterferon/ribavirin treatment period as prescribed by treating physician (e.g. 24 or 48 weeks) and treatment-free follow-up period of 24 weeks.

SUMMARY:
This observational study will assess predictors of early on-treatment and sustained virological response in treatment-naïve patients with chronic hepatitis C initiated on treatment with Pegasys (peginterferon alfa-2a) and ribavirin. Data will be collected during the treatment period (24 or 48 weeks) and 12 and 24 weeks after the end of treatment. Target sample size is <5000.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >/= 18 years of age
* chronic hepatitis C
* informed consent to data collection

Exclusion Criteria:

* co-infection with HIV or Hepatitis B Virus (HBV)
* previous treatment with peginterferon and/or ribavirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving peginterferon alfa-2a treatment at a medical centre
Sampling Method: Probability Sample
Enrollment: 4680 (Actual)
Dates: Start 2007-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (197):
- Austria (5):
  - Gratwein
  - Graz
  - Innsbruck
  - Linz
  - Vienna
- Brazil (13):
  - Salvador, Estado de Bahia
  - Goiânia, Goiás
  - Belo Horizonte, Minas Gerais
  - Belém, Pará
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Rio Grande, Rio Grande do Sul
  - Botucatu, São Paulo
  - Campinas, São Paulo
  - Ribeirão Preto, São Paulo
  - Santos, São Paulo
  - São Paulo, São Paulo
- Canada (29):
  - Calgary, Alberta
  - Edmonton, Alberta
  - Kelowna, British Columbia
  - Nanaimo, British Columbia
  - New Westminster, British Columbia
  - Prince George, British Columbia
  - Vancouver, British Columbia
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - St. John's, Newfoundland and Labrador
  - Barrie, Ontario
  - Brampton, Ontario
  - Etobicoke, Ontario
  - Greater Sudbury, Ontario
  - Guelph, Ontario
  - London, Ontario
  - Newmarket, Ontario
  - North Bay, Ontario
  - Oakville, Ontario
  - Oshawa, Ontario
  - Ottawa, Ontario
  - Scarborough Village, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Lévis, Quebec
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Charles-Borromée, Quebec
  - Saint-Jean-sur-Richelieu, Quebec
- Croatia (5):
  - Osijek
  - Pula
  - Split
  - Zadar
  - Zagreb
- France (88):
  - Agen
  - Aix-en-Provence
  - Albi
  - Amiens
  - Angers
  - Annecy
  - Antibes
  - Argenteuil
  - Aulnay-sous-Bois
  - Bastia
  - Beaumont
  - Beausoleil
  - Beauvais
  - Besançon
  - Béziers
  - Bordeaux
  - Boulogne-Billancourt
  - Bourgoin
  - Caen
  - Chambéry
  - Clermont-Ferrand
  - Clichy
  - Colmar
  - Cornebarrieu
  - Creil
  - Créteil
  - Dijon
  - Druex
  - Évreux
  - Freyming-Merlebach
  - Fréjus
  - Grasse
  - Grenoble
  - Hérouville-Saint-Clair
  - Hyères
  - La Rochelle
  - La Valette-du-Var
  - Lagny-sur-Marne
  - Le Chesnay
  - Le Havre
  - Le Kremlin-Bicêtre
  - Lille
  - Limoges
  - Lomme
  - Lorient
  - Lyon
  - Marseille
  - Martigues
  - Meaux
  - Melun
  - Menton
  - Metz
  - Monaco
  - Montauban
  - Montpellier
  - Mulhouse
  - Muret
  - Nanterre
  - Nantes
  - Nice
  - Nîmes
  - Ollioules
  - Orange
  - Orléans
  - Paris
  - Perpignan
  - Pessac
  - Périgueux
  - Poissy
  - Poitiers
  - Pont-à-Mousson
  - Reims
  - Rennes
  - Rouen
  - Saint-Dizier
  - Saint-Jean-de-Verges
  - Saint-Laurent-du-Var
  - Saint-Mandé
  - Sète
  - Ste Maxime
  - Strasbourg
  - Tarbes
  - Toulon
  - Toulouse
  - Tourcoing
  - Valenciennes
  - Vandœuvre-lès-Nancy
  - Villejuif
- Hungary (20):
  - Ajka
  - Békéscsaba
  - Budapest
  - Debrecen
  - Eger
  - Győr
  - Gyula
  - Kaposvár
  - Kecskemét
  - Kistarcsa
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Szeged
  - Szekszárd
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Tatabánya
  - Zalaegerszeg
- Mexico (8):
  - Chihuahua City
  - Culiacán
  - Guadalajara
  - Hermosillo
  - Mexicali
  - Mexico City
  - Monterrey
  - Puebla City
- Morocco (2):
  - Casablanca
  - Rabat
- Skopje, North Macedonia
- Poland (4):
  - Bydgoszcz
  - Lodz
  - Warsaw
  - Wroclaw
- Romania (9):
  - Arad
  - Brasov
  - Bucharest
  - Cluj-Napoca
  - Constanța
  - Iași
  - Sector 2
  - Târgu Mureş
  - Timișoara
- Serbia (3):
  - Belgrade
  - Niš
  - Novi Sad
- Slovenia (4):
  - Celje
  - Ljubljana
  - Maribor
  - Novo Mesto
- Sweden (6):
  - Eskilstuna
  - Halmstad
  - Huddinge
  - Linköping
  - Lund
  - Örebro

REFERENCES:
- [Derived] Ascione A, Bruno S, Coppola C, Mangia A, Orlandini A, Schmitz M, Deodato B, Puoti M. Treatment Outcomes and Predictors of Response in Treatment-Naive HCV Patients Treated with Peginterferon Alfa/Ribavirin in Real-World Italian Clinics: Sub-Analysis from the PROPHESYS Cohort. Hepatogastroenterology. 2014 Jun;61(132):1094-106. PMID 26158171
- [Derived] Ferenci P, Aires R, Ancuta I, Arohnson A, Cheinquer H, Delic D, Gschwantler M, Larrey D, Tallarico L, Schmitz M, Tatsch F, Ouzan D. A tool for selecting patients with a high probability of sustained virological response to peginterferon alfa-2a (40kD)/ribavirin. Liver Int. 2014 Nov;34(10):1550-9. doi: 10.1111/liv.12439. Epub 2014 Jan 9. PMID 24329937

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 4680 participants were enrolled into the study conducted from June 2007 to July 2011 at 332 centers in 14 countries.
Groups:
- Genotype 1: Eligible participants infected with hepatitis C virus (HCV) of Genotype 1 who received PEGASYS® (Pegylated Interferon [PEG-IFN]) alfa-2a plus ribavirin according to the standard of care and in line with summary of product characteristics (SPCs)/local labelling were observed for up to 72 weeks.
- Genotype 2: Eligible participants infected with HCV of Genotype 2 who received PEG-IFN alfa-2a plus ribavirin dose according to the standard of care and in line with SPCs/local labelling were observed for up to 72 weeks.
- Genotype 3: Eligible participants infected with HCV of Genotype 3 who received peginterferon alfa-2a plus ribavirin according to the standard of care and in line with SPCs/local labeling were observed for up to 72 weeks.
- Genotype 4: Eligible participants infected with HCV of Genotype 4 who received peginterferon alfa-2a plus ribavirin according to the standard of care and in line with SPCs/local labeling were observed for up to 72 weeks.
- Genotype 5/6: Eligible participants infected with HCV of Genotype 5/6 who received peginterferon alfa-2a plus ribavirin according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Genotype Unknown: Eligible participants infected with HCV of Genotype unknown who received PEG-IFN alfa-2a plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
Period: Overall Study
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Started | 3356 | 316 | 744 | 201 | 21 | 42
Completed | 2071 | 254 | 528 | 124 | 20 | 35
Not Completed | 1285 | 62 | 216 | 77 | 1 | 7
Not completed — Adverse Event | 43 | 1 | 3 | 0 | 0 | 0
Not completed — Death | 20 | 4 | 3 | 0 | 0 | 0
Not completed — Not meeting inclusion/exclusion criteria | 2 | 1 | 1 | 0 | 0 | 0
Not completed — Early termination | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Failed to return | 450 | 33 | 144 | 40 | 1 | 2
Not completed — Incomplete treatment | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lab test not done | 22 | 3 | 4 | 1 | 0 | 1
Not completed — Lack of Efficacy | 65 | 1 | 5 | 5 | 0 | 1
Not completed — Miscellaneous | 12 | 2 | 3 | 1 | 0 | 0
Not completed — New treatment started | 3 | 1 | 0 | 2 | 0 | 0
Not completed — Non-responders | 493 | 4 | 21 | 20 | 0 | 2
Not completed — Not categorized | 33 | 2 | 6 | 1 | 0 | 1
Not completed — Protocol Violation | 15 | 1 | 1 | 1 | 0 | 0
Not completed — Relapse | 44 | 5 | 14 | 4 | 0 | 0
Not completed — Result not available | 3 | 1 | 3 | 0 | 0 | 0
Not completed — Screen failure | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor decision | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment duration shortened | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment interrupted | 7 | 0 | 1 | 1 | 0 | 0
Not completed — Treatment not started | 14 | 2 | 4 | 0 | 0 | 0
Not completed — Treatment restarted | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Treatment stopped | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment unavailable | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment was stopped early | 7 | 0 | 0 | 0 | 0 | 0
Not completed — Other | 5 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 35 | 0 | 3 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled population included every participant for whom there was any data available in the PROPHESYS 1 database.
Groups:
- Genotype 1: Eligible participants infected with HCV of Genotype 1 who received PEG-IFN alfa-2a plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Genotype 2: Eligible participants infected with HCV of Genotype 2 who received PEG-IFN alfa-2a plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Genotype 3: Eligible participants infected with HCV of Genotype 3 who received PEG-IFN alfa-2a plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Genotype 4: Eligible participants infected with HCV of Genotype 4 who received PEG-IFN alfa-2a plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Genotype 5/6: Eligible participants infected with HCV of Genotype 5/6 who received PEG-IFN alfa-2a plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Genotype Unknown: Eligible participants infected with HCV of Unknown Genotype who received PEG-IFN alfa-2a plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
- Total: Total of all reporting groups
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown | Total
Number analyzed (Participants) | 3356 | 316 | 744 | 201 | 21 | 42 | 4680
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.1 (11.87) | 52.0 (11.74) | 40.8 (10.25) | 43.1 (9.87) | 52.5 (11.81) | 44.9 (10.62) | 46.3 (11.86)
Sex/Gender, Customized [Number; unit: Participants]
  Female | 1610 | 155 | 243 | 54 | 4 | 16 | 2082
  Male | 1746 | 161 | 501 | 147 | 17 | 25 | 2597
  Unknown | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virological Response by Genotype in Modified All Treated Population
Description: Sustained virological response (SVR) was defined as virological response (VR) at 24 weeks after end of treatment (EOT). Virological response was defined as hepatitis C virus ribonucleic acid (HCV RNA) of <15 international units per milliliter (IU/mL) as assessed by COBAS AmpliPrep/COBAS TaqMan (CAP/CTM) or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (lower limit of detection [LLOD] 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The SVR is reported in treatment naive hepatitis C virus (HCV) mono-infected modified all-treated (mTRT) who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The mTRT population included all participants who received at least one dose of peginterferon alfa-2a and ribavirin, and had at least one post-baseline HCV RNA test result. Participants with a baseline test result <50 IU/mL were excluded from the mTRT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Genotype 1: Eligible participants infected with HCV of Genotype 1 who received Peginterferon (PEG-IFN) alfa-2a plus ribavirin dose according to the standard of care and in line with SPCs/local labeling for up to 72 weeks were observed.
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2981 | 275 | 665 | 175 | 14 | 9
Percentage of participants | 40.6 [38.8 to 42.4] | 60.4 [54.3 to 66.2] | 55.0 [51.2 to 58.9] | 36.0 [28.9 to 43.6] | 57.1 [28.9 to 82.3] | 44.4 [13.7 to 78.8]

2. Primary Outcome: Percentage of Participants With Sustained Virological Response by Genotype in Per-Protocol Population
Description: Sustained virological response was defined as VR at 24 weeks after EOT. Virological response was defined as HCV RNA of <15 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The SVR is reported in treatment naive HCV mono-infected per protocol (PP) population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2554 | 234 | 597 | 152 | 12 | 7
Percentage of participants | 41.7 [39.8 to 43.7] | 62.0 [55.4 to 68.2] | 57.1 [53.0 to 61.1] | 38.8 [31.0 to 47.0] | 66.7 [34.9 to 90.1] | 42.9 [9.9 to 81.6]

3. Primary Outcome: Percentage of Participants With Modified Sustained Virological Response by Genotype in Modified All-Treated Population
Description: Modified sustained virological response (mSVR) was defined as modified virological response (mVR) of HCV RNA <50 IU/mL at 24 weeks after EOT. The mSVR is reported in treatment naive HCV mono-infected mTRT who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The mTRT population included all participants who received at least one dose of PEG-IFN alfa-2a and ribavirin, and had at least one post-baseline HCV RNA test result. Participants with a baseline test result of <50 IU/mL were excluded from the mTRT population.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2981 | 275 | 665 | 175 | 14 | 9
Percentage of participants | 43.2 [41.4 to 45.0] | 72.4 [66.7 to 77.6] | 60.5 [56.6 to 64.2] | 40.6 [33.2 to 48.2] | 71.4 [41.9 to 91.6] | 44.4 [13.7 to 78.8]
Statistical Analysis 1: Comparison: Genotype 1; The statistical analysis is presented for age per 10 years. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0126, Regression, Logistic; Odds Ratio (OR) = 0.903, 95% CI 2-sided [0.833 to 0.978]
Statistical Analysis 2: Comparison: Genotype 1; The statistical analysis is presented for Body Mass Index (BMI) in kilogram per square meter (kg/m^2). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0042, Regression, Logistic; Odds Ratio (OR) = 0.966, 95% CI 2-sided [0.944 to 0.989]
Statistical Analysis 3: Comparison: Genotype 1; The statistical analysis is presented for HCV RNA at Baseline (BL) in log10(IU/mL). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.732, 95% CI 2-sided [0.656 to 0.816]
Statistical Analysis 4: Comparison: Genotype 1; The statistical analysis is presented for liver fibrosis (no cirrhosis vs cirrhosis). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.686, 95% CI 2-sided [1.347 to 2.109]
Statistical Analysis 5: Comparison: Genotype 1; The statistical analysis is presented for liver fibrosis (not assessed/missed vs cirrhosis). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.4759, Regression, Logistic; Odds Ratio (OR) = 1.103, 95% CI 2-sided [0.843 to 1.442]
Statistical Analysis 6: Comparison: Genotype 1; The statistical analysis is presented for Alanine transaminase (ALT) ratio at BL (<=1 vs > 3). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0180, Regression, Logistic; Odds Ratio (OR) = 0.656, 95% CI 2-sided [0.462 to 0.930]
Statistical Analysis 7: Comparison: Genotype 1; The statistical analysis is presented for ALT ratio at BL (> 1 - 3 vs > 3). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0262, Regression, Logistic; Odds Ratio (OR) = 0.742, 95% CI 2-sided [0.570 to 0.965]
Statistical Analysis 8: Comparison: Genotype 1; The statistical analysis is presented for aspartate aminotransferase (AST) ratio at BL (> 1.5 vs <=1.5). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0069, Regression, Logistic; Odds Ratio (OR) = 0.717, 95% CI 2-sided [0.563 to 0.913]
Statistical Analysis 9: Comparison: Genotype 1; The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.062, 95% CI 2-sided [1.056 to 1.067]
Statistical Analysis 10: Comparison: Genotype 1; The statistical analysis is presented for cumulative ribavirin dose per 10000 mg, first 12 weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0062, Regression, Logistic; Odds Ratio (OR) = 1.107, 95% CI 2-sided [1.029 to 1.191]
Statistical Analysis 11: Comparison: Genotype 2; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0295, Regression, Logistic; Odds Ratio (OR) = 0.739, 95% CI 2-sided [0.563 to 0.970]
Statistical Analysis 12: Comparison: Genotype 2; The statistical analysis is presented for sex (male vs female). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.166, 95% CI 2-sided [0.083 to 0.329]
Statistical Analysis 13: Comparison: Genotype 2; [analysis description as in outcome 3, analysis 9]; Test type: Superiority or Other; p = 0.0048, Regression, Logistic; Odds Ratio (OR) = 1.049, 95% CI 2-sided [1.015 to 1.084]
Statistical Analysis 14: Comparison: Genotype 2; The statistical analysis is presented for cumulative PEG-IFN alfa-2a dose per 1000 ug, first 12 weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0019, Regression, Logistic; Odds Ratio (OR) = 7.797, 95% CI 2-sided [2.136 to 28.458]
Statistical Analysis 15: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 12]; Test type: Superiority or Other; p = 0.0255, Regression, Logistic; Odds Ratio (OR) = 0.638, 95% CI 2-sided [0.431 to 0.946]
Statistical Analysis 16: Comparison: Genotype 3; The statistical analysis is presented for HCV RNA at BL in log10(IU/mL). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0059, Regression, Logistic; Odds Ratio (OR) = 0.755, 95% CI 2-sided [0.618 to 0.922]
Statistical Analysis 17: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 2.521, 95% CI 2-sided [1.501 to 4.236]
Statistical Analysis 18: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 5]; Test type: Superiority or Other; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 2.602, 95% CI 2-sided [1.463 to 4.627]
Statistical Analysis 19: Comparison: Genotype 3; The statistical analysis is presented for mode of infection (other vs injection drug U). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0034, Regression, Logistic; Odds Ratio (OR) = 1.727, 95% CI 2-sided [1.198 to 2.491]
Statistical Analysis 20: Comparison: Genotype 3; The statistical analysis is presented for AST ratio at BL (> 1.5 vs <=1.5). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0014, Regression, Logistic; Odds Ratio (OR) = 0.545, 95% CI 2-sided [0.376 to 0.792]
Statistical Analysis 21: Comparison: Genotype 3; The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.047, 95% CI 2-sided [1.029 to 1.065]
Statistical Analysis 22: Comparison: Genotype 1; The statistical analysis is presented for age per 10 years. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0074, Regression, Logistic; Odds Ratio (OR) = 0.896, 95% CI 2-sided [0.827 to 0.971]
Statistical Analysis 23: Comparison: Genotype 1; The statistical analysis is presented for BMI in kg/m^2. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0088, Regression, Logistic; Odds Ratio (OR) = 0.971, 95% CI 2-sided [0.950 to 0.993]
Statistical Analysis 24: Comparison: Genotype 1; The statistical analysis is presented for HCV RNA at BL in log10(IU/mL). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.719, 95% CI 2-sided [0.643 to 0.803]
Statistical Analysis 25: Comparison: Genotype 1; The statistical analysis is presented for liver fibrosis (no cirrhosis vs cirrhosis). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.683, 95% CI 2-sided [1.346 to 2.106]
Statistical Analysis 26: Comparison: Genotype 1; The statistical analysis is presented for liver fibrosis (not assessed/missing vs cirrhosis). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.4479, Regression, Logistic; Odds Ratio (OR) = 1.110, 95% CI 2-sided [0.848 to 1.453]
Statistical Analysis 27: Comparison: Genotype 1; The statistical analysis is presented for ALT ratio at BL (<=1 vs > 3). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0123, Regression, Logistic; Odds Ratio (OR) = 0.640, 95% CI 2-sided [0.451 to 0.908]
Statistical Analysis 28: Comparison: Genotype 1; The statistical analysis is presented for ALT ratio at BL (> 1 - 3 vs > 3). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0147, Regression, Logistic; Odds Ratio (OR) = 0.720, 95% CI 2-sided [0.553 to 0.937]
Statistical Analysis 29: Comparison: Genotype 1; The statistical analysis is presented for AST ratio at BL (> 1.5 vs <=1.5). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0071, Regression, Logistic; Odds Ratio (OR) = 0.718, 95% CI 2-sided [0.564 to 0.914]
Statistical Analysis 30: Comparison: Genotype 1; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.058, 95% CI 2-sided [1.052 to 1.064]
Statistical Analysis 31: Comparison: Genotype 1; The statistical analysis is presented for cumulative ribavirin dose per 10000 mg. The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0019, Regression, Logistic; Odds Ratio (OR) = 1.014, 95% CI 2-sided [1.005 to 1.023]
Statistical Analysis 32: Comparison: Genotype 2; [analysis description as in outcome 3, analysis 22]; Test type: Superiority or Other; p = 0.0083, Regression, Logistic; Odds Ratio (OR) = 0.701, 95% CI 2-sided [0.539 to 0.913]
Statistical Analysis 33: Comparison: Genotype 2; The statistical analysis is presented for sex (male vs female). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.174, 95% CI 2-sided [0.090 to 0.338]
Statistical Analysis 34: Comparison: Genotype 2; [analysis description as in outcome 3, analysis 21]; Test type: Superiority or Other; p = 0.0008, Regression, Logistic; Odds Ratio (OR) = 1.057, 95% CI 2-sided [1.023 to 1.091]
Statistical Analysis 35: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 33]; Test type: Superiority or Other; p = 0.0255, Regression, Logistic; Odds Ratio (OR) = 0.638, 95% CI 2-sided [0.431 to 0.946]
Statistical Analysis 36: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 24]; Test type: Superiority or Other; p = 0.0059, Regression, Logistic; Odds Ratio (OR) = 0.755, 95% CI 2-sided [0.618 to 0.922]
Statistical Analysis 37: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 25]; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 2.521, 95% CI 2-sided [1.501 to 4.236]
Statistical Analysis 38: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 26]; Test type: Superiority or Other; p = 0.0011, Regression, Logistic; Odds Ratio (OR) = 2.602, 95% CI 2-sided [1.463 to 4.627]
Statistical Analysis 39: Comparison: Genotype 3; The statistical analysis is presented for mode of infection (other vs injection drug U). The logistic regression analysis for mSVR was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0034, Regression, Logistic; Odds Ratio (OR) = 1.727, 95% CI 2-sided [1.198 to 2.491]
Statistical Analysis 40: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 29]; Test type: Superiority or Other; p = 0.0014, Regression, Logistic; Odds Ratio (OR) = 0.545, 95% CI 2-sided [0.376 to 0.792]
Statistical Analysis 41: Comparison: Genotype 1; The statistical analysis is presented for age per 10 years. The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0042, Regression, Logistic; Odds Ratio (OR) = 0.890, 95% CI 2-sided [0.822 to 0.964]
Statistical Analysis 42: Comparison: Genotype 1; The statistical analysis is presented for sex (male vs female). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0363, Regression, Logistic; Odds Ratio (OR) = 0.824, 95% CI 2-sided [0.687 to 0.988]
Statistical Analysis 43: Comparison: Genotype 1; The statistical analysis is presented for HCV RNA at BL in log10(IU/mL). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 0.842, 95% CI 2-sided [0.751 to 0.944]
Statistical Analysis 44: Comparison: Genotype 1; The statistical analysis is presented for liver fibrosis (no cirrhosis vs cirrhosis). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 1.477, 95% CI 2-sided [1.183 to 1.844]
Statistical Analysis 45: Comparison: Genotype 1; The statistical analysis is presented for liver fibrosis (not assessed/missing vs cirrhosis). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.3810, Regression, Logistic; Odds Ratio (OR) = 1.128, 95% CI 2-sided [0.862 to 1.477]
Statistical Analysis 46: Comparison: Genotype 1; The statistical analysis is presented for AST ratio at BL (> 1.5 vs <=1.5). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0279, Regression, Logistic; Odds Ratio (OR) = 0.812, 95% CI 2-sided [0.674 to 0.978]
Statistical Analysis 47: Comparison: Genotype 1; The statistical analysis is presented for On-treatment response (RVR vs no RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 45.894, 95% CI 2-sided [27.972 to 75.299]
Statistical Analysis 48: Comparison: Genotype 1; The statistical analysis is presented for on-treatment response (cEVR vs no RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 32.176, 95% CI 2-sided [20.129 to 51.434]
Statistical Analysis 49: Comparison: Genotype 1; The statistical analysis is presented for on-treatment response (pEVR vs NO RVR/EVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 6.928, 95% CI 2-sided [4.291 to 11.188]
Statistical Analysis 50: Comparison: Genotype 2; [analysis description as in outcome 3, analysis 41]; Test type: Superiority or Other; p = 0.0204, Regression, Logistic; Odds Ratio (OR) = 0.733, 95% CI 2-sided [0.564 to 0.953]
Statistical Analysis 51: Comparison: Genotype 2; [analysis description as in outcome 3, analysis 42]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.170, 95% CI 2-sided [0.087 to 0.331]
Statistical Analysis 52: Comparison: Genotype 2; The statistical analysis is presented for on-treatment response, combined (RVR vs no RVR). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 2.806, 95% CI 2-sided [1.514 to 5.201]
Statistical Analysis 53: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 42]; Test type: Superiority or Other; p = 0.0459, Regression, Logistic; Odds Ratio (OR) = 0.663, 95% CI 2-sided [0.443 to 0.993]
Statistical Analysis 54: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 43]; Test type: Superiority or Other; p = 0.0087, Regression, Logistic; Odds Ratio (OR) = 0.758, 95% CI 2-sided [0.616 to 0.932]
Statistical Analysis 55: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 44]; Test type: Superiority or Other; p = 0.0064, Regression, Logistic; Odds Ratio (OR) = 2.054, 95% CI 2-sided [1.224 to 3.447]
Statistical Analysis 56: Comparison: Genotype 3; The statistical analysis is presented for liver fibrosis (not assessed/missed vs cirrhosis). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0271, Regression, Logistic; Odds Ratio (OR) = 1.931, 95% CI 2-sided [1.077 to 3.461]
Statistical Analysis 57: Comparison: Genotype 3; The statistical analysis is presented for mode of infection (other vs injection drug U). The logistic regression analysis for mSVR was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0039, Regression, Logistic; Odds Ratio (OR) = 1.738, 95% CI 2-sided [1.194 to 2.528]
Statistical Analysis 58: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 46]; Test type: Superiority or Other; p = 0.0035, Regression, Logistic; Odds Ratio (OR) = 0.565, 95% CI 2-sided [0.386 to 0.829]
Statistical Analysis 59: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 47]; Test type: Superiority or Other; p = 0.0071, Regression, Logistic; Odds Ratio (OR) = 5.533, 95% CI 2-sided [1.593 to 19.219]
Statistical Analysis 60: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 48]; Test type: Superiority or Other; p = 0.3042, Regression, Logistic; Odds Ratio (OR) = 1.964, 95% CI 2-sided [0.542 to 7.114]
Statistical Analysis 61: Comparison: Genotype 3; [analysis description as in outcome 3, analysis 49]; Test type: Superiority or Other; p = 0.4100, Regression, Logistic; Odds Ratio (OR) = 1.726, 95% CI 2-sided [0.471 to 6.318]

4. Primary Outcome: Percentage of Participants With Modified Sustained Virological Response by Genotype in Per-Protocol Population
Description: Modified sustained virological response is defined as mVR of HCV RNA <50 IU/mL at 24 weeks after EOT. The mSVR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2554 | 234 | 597 | 152 | 12 | 7
Percentage of participants | 44.4 [42.5 to 46.4] | 74.4 [68.3 to 79.8] | 62.3 [58.3 to 66.2] | 44.1 [36.0 to 52.4] | 83.3 [51.6 to 97.9] | 42.9 [9.9 to 81.6]

5. Primary Outcome: Percentage of Participants With Predictive Values of Virological Response by Week 4 and Week 12 on Modified Sustained Virological Response by Genotype After Treatment Initiation in Modified All-Treated Population
Description: The probability that a participant who developed VR by Week 4 and 12 and also achieved mSVR at 24 weeks after EOT was called the positive predictive value (PPV) of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 4 and 12 and also failed to achieve mSVR at 24 weeks after EOT was called the negative predictive value (NPV) of the VR by Wk 4 and 12 for mSVR. Predictive values of VR are reported in treatment naive HCV mono-infected mTRT participants who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The mTRT population included all participants who received at least one dose of PEG-IFN alfa-2a and ribavirin, and had at least one post-baseline HCV RNA test result. Participants with a baseline test result <50 IU/mL were excluded from the mTRT population. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2957 | 272 | 652 | 173 | 14 | 8
Percentage of participants
  Week 4, PPV (n=2802, 263, 618, 159, 12, 8) | 71.4 [67.6 to 75.0] | 77.3 [70.3 to 83.4] | 71.1 [66.4 to 75.6] | 68.6 [54.1 to 80.9] | 75.0 [19.4 to 99.4] | 100.0 [15.8 to 100.0]
  Week 4, NPV (n=2802, 263, 618, 159, 12, 8) | 64.1 [62.1 to 66.1] | 34.1 [24.5 to 44.7] | 55.6 [48.8 to 62.2] | 70.4 [60.8 to 78.8] | 37.5 [8.5 to 75.5] | 66.7 [22.3 to 95.7]
  Week12, PPV (n=2957, 272, 652, 173, 14, 8) | 65.3 [62.9 to 67.7] | 74.5 [68.1 to 80.2] | 65.8 [61.5 to 69.9] | 52.7 [43.0 to 62.3] | 80.0 [44.4 to 97.5] | 100.0 [39.8 to 100.0]
  Week 12, NPV (n=2957, 272, 652, 173, 14, 8) | 82.4 [80.3 to 84.4] | 33.3 [21.7 to 46.7] | 58.0 [49.3 to 66.3] | 81.0 [69.1 to 89.8] | 50.0 [6.8 to 93.2] | 100.0 [39.8 to 100.0]

6. Primary Outcome: Percentage of Participants With Predictive Values of Virological Response by Week 4 and 12 on Modified Sustained Virological Response by Genotype After Treatment Initiation in Per-Protocol Population
Description: The probability that a participant who developed VR by Week 4 and 12 and also achieved mSVR at 24 weeks after EOT was called the PPV of the VR by Wk 4 for mSVR. The probability that a participant who failed to develop VR by Wk 4 and 12 and also failed to achieve mSVR at 24 weeks after EOT was called the NPV of the VR by Wk 4 and 12 for mSVR. Predictive values of VR are reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The PP population included all participants who met the inclusion/exclusion criteria. n = the number of participants analyzed at a given time point.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2535 | 231 | 586 | 150 | 12 | 6
Percentage of participants
  Week 4, PPV (n=2408, 222, 556, 139, 10, 6) | 72.2 [68.0 to 76.1] | 79.2 [71.8 to 85.4] | 73.2 [68.3 to 77.7] | 67.3 [52.5 to 80.1] | 75.0 [19.4 to 99.4] | 100.0 [15.8 to 100.0]
  Week 4, NPV (n=2408, 222, 556, 139, 10, 6) | 63.0 [60.8 to 65.2] | 31.5 [21.1 to 43.4] | 55.1 [47.8 to 62.1] | 66.7 [55.9 to 76.3] | 16.7 [0.4 to 64.1] | 75.0 [19.4 to 99.4]
  Week 12, PPV (n=2535, 231, 586, 150, 12, 6) | 66.9 [64.4 to 69.4] | 76.7 [69.8 to 82.6] | 67.3 [62.9 to 71.5] | 56.1 [45.7 to 66.1] | 88.9 [51.8 to 99.7] | 100.0 [29.2 to 100.0]
  Week 12, NPV (n=2535, 231, 586, 150, 12, 6) | 81.6 [79.3 to 83.8] | 31.4 [19.1 to 45.9] | 55.9 [46.5 to 65.1] | 78.8 [65.3 to 88.9] | 33.3 [0.8 to 90.6] | 100.0 [29.2 to 100.0]

7. Secondary Outcome: Percentage of Participants With Virological Response by Genotype in Modified All-Treated Population Over Time
Description: Virological response was defined as HCV RNA <15 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The VR is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At Week 2, Week 4, and Week 12, EOT, and 12 weeks after EOT
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2981 | 275 | 665 | 175 | 14 | 9
Percentage of participants
  At Week 2 | 4.8 [4.1 to 5.6] | 24.7 [19.7 to 30.3] | 16.2 [13.5 to 19.3] | 8.6 [4.9 to 13.7] | 14.3 [1.8 to 42.8] | 11.1 [0.3 to 48.2]
  At Week 4 | 19.7 [18.3 to 21.2] | 62.5 [56.5 to 68.3] | 59.4 [55.6 to 63.2] | 29.1 [22.5 to 36.5] | 28.6 [8.4 to 58.1] | 22.2 [2.8 to 60.0]
  At Week 12 | 53.2 [51.4 to 55.0] | 77.1 [71.7 to 81.9] | 77.3 [73.9 to 80.4] | 62.9 [55.2 to 70.0] | 71.4 [41.9 to 91.6] | 44.4 [13.7 to 78.8]
  At EOT | 62.1 [60.4 to 63.9] | 75.6 [70.1 to 80.6] | 78.0 [74.7 to 81.1] | 59.4 [51.8 to 66.8] | 71.4 [41.9 to 91.6] | 44.4 [13.7 to 78.8]
  At 12 Weeks after EOT | 43.2 [41.5 to 45.0] | 64.0 [58.0 to 69.7] | 59.5 [55.7 to 63.3] | 40.6 [33.2 to 48.2] | 57.1 [28.9 to 82.3] | 44.4 [13.7 to 78.8]

8. Secondary Outcome: Percentage of Participants With Virological Response by Genotype in Per-Protocol Population Over Time
Description: Virological response was defined as HCV RNA <15 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The VR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At Week 2, Week 4, Week 12, EOT, and 12 weeks after EOT
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2554 | 234 | 597 | 152 | 12 | 7
Percentage of participants
  At Week 2 | 4.8 [4.0 to 5.7] | 26.1 [20.6 to 32.2] | 16.8 [13.8 to 20.0] | 8.6 [4.6 to 14.2] | 16.7 [2.1 to 48.4] | 14.3 [0.4 to 57.9]
  At Week 4 | 19.6 [18.1 to 21.2] | 63.7 [57.2 to 69.8] | 60.0 [55.9 to 63.9] | 32.2 [24.9 to 40.3] | 33.3 [9.9 to 65.1] | 28.6 [3.7 to 71.0]
  At Week 12 | 53.2 [51.2 to 55.1] | 76.9 [71.0 to 82.2] | 78.4 [74.9 to 81.6] | 64.5 [56.3 to 72.1] | 75.0 [42.8 to 94.5] | 42.9 [9.9 to 81.6]
  At EOT | 62.5 [60.6 to 64.4] | 76.1 [70.1 to 81.4] | 79.6 [76.1 to 82.7] | 61.8 [53.6 to 69.6] | 75.0 [42.8 to 94.5] | 42.9 [9.9 to 81.6]
  At 12 weeks after EOT | 44.2 [42.3 to 46.2] | 65.8 [59.3 to 71.9] | 61.8 [57.8 to 65.7] | 43.4 [35.4 to 51.7] | 66.7 [34.9 to 90.1] | 42.9 [9.9 to 81.6]

9. Secondary Outcome: Percentage of Participants With Modified Virological Response by Genotype in Modified All-Treated Population Over Time
Description: Modified virological response was defined as HCV RNA <50 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The mVR is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At Week 2, Week 4, Week 12, EOT, and 12 weeks after EOT
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2981 | 275 | 665 | 175 | 14 | 9
Percentage of participants
  At Week 2 | 6.7 [5.8 to 7.6] | 31.3 [25.8 to 37.1] | 23.0 [19.9 to 26.4] | 13.7 [9.0 to 19.7] | 28.6 [8.4 to 58.1] | 11.1 [0.3 to 48.2]
  At Week 4 | 25.9 [24.4 to 27.5] | 82.5 [77.5 to 86.8] | 73.2 [69.7 to 76.6] | 39.4 [32.1 to 47.1] | 50.0 [23.0 to 77.0] | 33.3 [7.5 to 70.1]
  At Week 12 | 62.3 [60.6 to 64.1] | 96.0 [93.0 to 98.0] | 93.1 [90.9 to 94.9] | 73.1 [65.9 to 79.6] | 100.0 [76.8 to 100.0] | 44.4 [13.7 to 78.8]
  At EOT | 67.7 [65.9 to 69.3] | 92.4 [88.6 to 95.2] | 88.7 [86.1 to 91.0] | 68.6 [61.1 to 75.4] | 92.9 [66.1 to 99.8] | 55.6 [21.2 to 86.3]
  At 12 weeks after EOT | 46.2 [44.4 to 48.0] | 76.4 [70.9 to 81.3] | 65.0 [61.2 to 68.6] | 46.3 [38.7 to 54.0] | 85.7 [57.2 to 98.2] | 44.4 [13.7 to 78.8]

10. Secondary Outcome: Percentage of Participants With Modified Virological Response by Genotype in Per-Protocol Population Over Time
Description: Modified virological response is defined as HCV RNA <50 IU/mL as assessed by CAP/CTM or another HCV RNA test with at least the same degree of sensitivity. The CAP/CTM test is an in vitro nucleic acid amplification test for the quantification of HCV. This test possesses a high sensitivity (LLOD 15 IU/mL) and a broad linear range of quantification (43 IU/mL up to 69 million IU/mL) in all HCV genotypes. The mVR is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At Week 2, Week 4, Week 12, EOT, and 12 weeks after EOT
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2554 | 234 | 597 | 152 | 12 | 7
Percentage of participants
  At Week 2 | 6.6 [5.7 to 7.7] | 32.5 [26.5 to 38.9] | 23.6 [20.3 to 27.2] | 13.8 [8.8 to 20.3] | 33.3 [9.9 to 65.1] | 14.3 [0.4 to 57.9]
  At Week 4 | 25.7 [24.0 to 27.5] | 81.6 [76.1 to 86.4] | 73.4 [69.6 to 76.9] | 42.1 [34.2 to 50.4] | 58.3 [27.7 to 84.8] | 42.9 [9.9 to 81.6]
  At Week 12 | 62.5 [60.5 to 64.3] | 95.3 [91.7 to 97.6] | 93.8 [91.6 to 95.6] | 74.3 [66.6 to 81.1] | 100.0 [73.5 to 100.0] | 42.9 [9.9 to 81.6]
  At EOT | 68.0 [66.2 to 69.8] | 92.7 [88.6 to 95.7] | 89.4 [86.7 to 91.8] | 71.7 [63.8 to 78.7] | 91.7 [61.5 to 99.8] | 42.9 [9.9 to 81.6]
  At 12 week after EOT | 47.3 [45.3 to 49.2] | 78.6 [72.8 to 83.7] | 67.0 [63.1 to 70.8] | 49.3 [41.1 to 57.6] | 91.7 [61.5 to 99.8] | 42.9 [9.9 to 81.6]

11. Secondary Outcome: Percentage of Participants With At Least 2-logarithm10 Drop in Hepatitis C Virus Deoxyribonucleic Acid by Genotype in Modified All-Treated Population at Week 2, Week 4 and Week 12
Description: Participants with 2-logarithm (log) drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 2 log drop in HCV RNA was defined as drop of HCV viral load by 99%. The 2 log drop in HCV RNA is reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a.
Time Frame: At Week 2, Week 4, and Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2981 | 275 | 665 | 175 | 14 | 9
Percentage of participants
  >=2-log10 drop at Week 2 | 21.5 [20.0 to 23.0] | 49.1 [43.0 to 55.2] | 40.6 [36.8 to 44.4] | 22.3 [16.4 to 29.2] | 42.9 [17.7 to 71.1] | 11.1 [0.3 to 48.2]
  >=2-log10 drop at Week 4 | 55.2 [53.4 to 57.0] | 92.4 [88.6 to 95.2] | 87.8 [85.1 to 90.2] | 56.0 [48.3 to 63.5] | 85.7 [57.2 to 98.2] | 44.4 [13.7 to 78.8]
  >=2-log10 drop at Week 12 | 81.8 [80.4 to 83.2] | 98.2 [95.8 to 99.4] | 95.6 [93.8 to 97.1] | 82.9 [76.4 to 88.1] | 100.0 [76.8 to 100.0] | 44.4 [13.7 to 78.8]

12. Secondary Outcome: Percentage of Participants With At Least a 2-logarithm10 Drop in Hepatitis C Virus Deoxyribonucleic Acid by Genotype in Per-Protocol Population at Week 2, Week 4 and Week 12
Description: Participants with 2-log drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 2 log drop in HCV RNA was defined as drop of HCV viral load by 99%. The 2 log drop in HCV RNA is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a.
Time Frame: Week 2, Week 4, and Week 12
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2554 | 234 | 597 | 152 | 12 | 7
Percentage of participants
  >=2-log 10 drop by Week 2 | 21.3 [19.7 to 22.9] | 49.1 [42.6 to 55.7] | 40.5 [36.6 to 44.6] | 22.4 [16.0 to 29.8] | 41.7 [15.2 to 72.3] | 14.3 [0.4 to 57.9]
  >=2-log 10 drop by Week 4 | 55.6 [53.6 to 57.5] | 91.0 [86.6 to 94.4] | 88.1 [85.2 to 90.6] | 59.9 [51.6 to 67.7] | 83.3 [51.6 to 97.9] | 42.9 [9.9 to 81.6]
  >=2-log 10 drop by Week 12 | 82.5 [81.0 to 84.0] | 97.9 [95.1 to 99.3] | 96.0 [94.1 to 97.4] | 84.2 [77.4 to 89.6] | 100.0 [73.5 to 100.0] | 42.9 [9.9 to 81.6]

13. Secondary Outcome: Percentage of Participants With At Least 1-logarithm10 Drop in Hepatitis C Virus Deoxyribonucleic Acid by Genotype in Modified All-Treated Population at Week 2, Week 4 and Week 12
Description: Participants with 1-log drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 1- log drop in HCV RNA was defined as drop of HCV viral load by 90%. The 1- log drop in HCV RNA was reported in treatment naive HCV mono-infected mTRT population who received PEG-IFN alfa-2a.
Time Frame: Week 2, Week 4, and Week 12
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2981 | 275 | 665 | 175 | 14 | 9
Percentage of participants
  >=1-log10 drop by Week 2 | 33.6 [31.9 to 35.3] | 51.6 [45.6 to 57.7] | 46.0 [42.2 to 49.9] | 35.4 [28.4 to 43.0] | 42.9 [17.7 to 71.1] | 11.1 [0.3 to 48.2]
  >=1-log10 drop by Week 4 | 75.0 [73.4 to 76.6] | 93.8 [90.3 to 96.4] | 90.2 [87.7 to 92.4] | 72.6 [65.3 to 79.0] | 85.7 [57.2 to 98.2] | 55.6 [21.2 to 86.3]
  >=1-log10 drop by Week 12 | 90.5 [89.4 to 91.5] | 98.5 [96.3 to 99.6] | 96.5 [94.9 to 97.8] | 90.9 [85.6 to 94.7] | 100.0 [76.8 to 100.0] | 66.7 [29.9 to 92.5]

14. Secondary Outcome: Percentage of Participants With At Least 1 Log Drop in Hepatitis C Virus Deoxyribonucleic Acid by Genotype in Per-Protocol Population at Week 2, Week 4 and Week 12
Description: Participants with 1-log drop in HCV RNA including HCV RNA values <50 IU/mL in the serum from baseline to Week 2, Week 4 and Week 12, expressed in terms of a logarithmic scale with base 10 were evaluated and reported. A 1- log drop in HCV RNA was defined as drop of HCV viral load by 90%. The 1- log drop in HCV RNA was reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a.
Time Frame: Week 2, Week 4, and Week 12
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2554 | 234 | 597 | 152 | 12 | 7
Percentage of participants
  >=1-log10 drop by Week 2 | 33.5 [31.7 to 35.4] | 51.7 [45.1 to 58.3] | 46.1 [42.0 to 50.2] | 35.5 [27.9 to 43.7] | 41.7 [15.2 to 72.3] | 14.3 [0.4 to 57.9]
  >=1-log10 drop by Week 4 | 76.3 [74.6 to 77.9] | 92.7 [88.6 to 95.7] | 90.6 [88.0 to 92.8] | 76.3 [68.7 to 82.8] | 83.3 [51.6 to 97.9] | 57.1 [18.4 to 90.1]
  >=1-log10 drop by Week 12 | 91.6 [90.5 to 92.7] | 98.3 [95.7 to 99.5] | 96.8 [95.1 to 98.1] | 92.1 [86.6 to 95.9] | 100.0 [73.5 to 100.0] | 71.4 [29.0 to 96.3]

15. Secondary Outcome: Number of Participants With Response by Disjoint Categories by Genotype in Modified All-Treated Population at Week 4 and Week 12
Description: Rapid virological response (RVR) was defined as VR by Week 4, Modified rapid virological response (mRVR) was defined as mVR by Week 4, Complete early virological response (cEVR) was defined as VR by Week 12, but no RVR, Modified complete early virological response (mcEVR) was defined as mVR by Week 12, but no mRVR, Partial early virological response (pEVR) was defined as at least a 2-log10 drop in HCV RNA as compared to baseline (including HCV RNA values <50 IU/mL) by, Week 12, but no RVR and no cEVR, Modified partial early virological response (mpEVR) was defined as at least a 2-log10 drop in HCV RNA as compared to baseline by Week 12, but no mRVR and no mcEVR. The data is reported in treatment naive HCV mono-infected mTRT participants who received PEG-IFN alfa-2a.
Time Frame: Week 4 and Week 12
Population: The mTRT population included all participants who received at least one dose of PEG-IFN alfa-2a and ribavirin, and had at least one post-baseline HCV RNA test result. Participants with a baseline test result <50 IU/mL were excluded from the mTRT population.
Measure: Number; unit: Participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2981 | 275 | 665 | 175 | 14 | 9
Participants
  RVR at Week 4 | 588 | 172 | 395 | 51 | 4 | 2
  mRVR at Week 4 | 773 | 227 | 487 | 69 | 7 | 3
  cEVR at Week 12 | 998 | 40 | 119 | 59 | 6 | 2
  mcEVR at Week 12 | 1085 | 37 | 132 | 59 | 7 | 1
  pEVR at Week 12 | 853 | 58 | 122 | 35 | 4 | 0
  mpEVR at Week 12 | 581 | 6 | 17 | 17 | 0 | 0

16. Secondary Outcome: Number of Participants With Response by Disjoint Categories by Genotype in Per-Protocol Population at Week 4 and Week 12
Description: RVR defined was as VR by Week 4, mRVR was defined as mVR by Week 4, cEVR was defined as VR by Week 12, but no RVR, mcEVR was defined as mVR by Week 12, but no mRVR, pEVR was defined as at least a 2-log10 drop in HCV RNA as compared to baseline (including HCV RNA values <50 IU/mL) by Week 12, but no RVR and no cEVR, mpEVR was defined as at least a 2-log10 drop in HCV RNA as compared to baseline by Week 12, but no mRVR and no mcEVR. The data is reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a.
Time Frame: At Week 4 and Week 12
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number; unit: Participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 2554 | 234 | 597 | 152 | 12 | 7
Participants
  RVR at Week 4 | 500 | 149 | 358 | 49 | 4 | 2
  mRVR at Week 4 | 657 | 191 | 438 | 64 | 7 | 3
  cEVR at Week 12 | 858 | 31 | 110 | 49 | 5 | 1
  mcEVR at Week 12 | 938 | 32 | 122 | 49 | 5 | 0
  pEVR at Week 12 | 749 | 49 | 105 | 30 | 3 | 0
  mpEVR at Week 12 | 512 | 6 | 13 | 15 | 0 | 0

17. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Modified All-Treated Population at 12 Weeks After End of Treatment
Description: Participants whose last test result in their respective follow-up time window showed mVR were considered to have maintained their modified end of treatment response (mEOT-R). Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. The percentage of participants with relapse is reported in treatment naive mTRT population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 12 Weeks after EOT
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 775 | 127 | 247 | 54 | 6 | 1
Percentage of participants | 26.5 | 10.2 | 19.4 | 29.6 | 0.0 | 0.0

18. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Per Protocol Population at 12 Weeks After End of Treatment
Description: Participants whose last test result in their respective follow-up time window showed mVR were considered to have maintained their mEOT-R. Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. The percentage of participants with relapse is reported in treatment naive PP population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 12 weeks after EOT
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number; unit: Percentage of Participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 671 | 116 | 234 | 49 | 5 | 1
Percentage of Participants | 24.4 | 10.3 | 18.4 | 28.6 | 0.0 | 0.0

19. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Modified All-Treated Population at 24 Weeks After End of Treatment
Description: Participants whose last test result in the follow-up time window showed mVR were considered to have maintained their mEOT-R. Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. The percentage of participants with relapse was reported in treatment naive mTRT population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 1751 | 227 | 487 | 95 | 11 | 4
Percentage of participants | 27.1 | 12.3 | 17.9 | 25.3 | 9.1 | 0.0
Statistical Analysis 1: Comparison: Genotype 1; The statistical analysis is presented for age per 10 years. The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.379, 95% CI 2-sided [1.236 to 1.538]
Statistical Analysis 2: Comparison: Genotype 1; The statistical analysis is presented for BMI in kg/m^2. The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0251, Regression, Logistic; Odds Ratio (OR) = 1.033, 95% CI 2-sided [1.004 to 1.063]
Statistical Analysis 3: Comparison: Genotype 1; The statistical analysis is presented for HCV RNA at BL in log10(IU/mL). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.585, 95% CI 2-sided [1.358 to 1.849]
Statistical Analysis 4: Comparison: Genotype 1; The statistical analysis is presented for ALT ratio at BL (<=1 vs > 3). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0317, Regression, Logistic; Odds Ratio (OR) = 1.501, 95% CI 2-sided [1.036 to 2.174]
Statistical Analysis 5: Comparison: Genotype 1; The statistical analysis is presented for ALT ratio at BL (> 1 - 3 vs > 3). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0129, Regression, Logistic; Odds Ratio (OR) = 1.493, 95% CI 2-sided [1.089 to 2.048]
Statistical Analysis 6: Comparison: Genotype 1; The statistical analysis is presented for Platelets x 10^9/L at BL (< 140 vs >=180). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0128, Regression, Logistic; Odds Ratio (OR) = 1.616, 95% CI 2-sided [1.107 to 2.357]
Statistical Analysis 7: Comparison: Genotype 1; The statistical analysis is presented for Platelets x 10^9/L at BL (>=140 - < 180 vs >=180). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.7809, Regression, Logistic; Odds Ratio (OR) = 1.046, 95% CI 2-sided [0.763 to 1.432]
Statistical Analysis 8: Comparison: Genotype 1; The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.969, 95% CI 2-sided [0.962 to 0.976]
Statistical Analysis 9: Comparison: Genotype 1; The statistical analysis is presented for Cumulative PEG-IFN alfa-2a dose per 1000 ug, first 12 weeks. The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0189, Regression, Logistic; Odds Ratio (OR) = 4.298, 95% CI 2-sided [1.273 to 14.512]
Statistical Analysis 10: Comparison: Genotype 2; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.0316, Regression, Logistic; Odds Ratio (OR) = 1.567, 95% CI 2-sided [1.040 to 2.359]
Statistical Analysis 11: Comparison: Genotype 2; The statistical analysis is presented for sex (male vs female). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0024, Regression, Logistic; Odds Ratio (OR) = 4.495, 95% CI 2-sided [1.701 to 11.879]
Statistical Analysis 12: Comparison: Genotype 2; [analysis description as in outcome 19, analysis 2]; Test type: Superiority or Other; p = 0.0247, Regression, Logistic; Odds Ratio (OR) = 1.112, 95% CI 2-sided [1.014 to 1.219]
Statistical Analysis 13: Comparison: Genotype 2; [analysis description as in outcome 19, analysis 3]; Test type: Superiority or Other; p = 0.0258, Regression, Logistic; Odds Ratio (OR) = 1.844, 95% CI 2-sided [1.077 to 3.158]
Statistical Analysis 14: Comparison: Genotype 3; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 1.677, 95% CI 2-sided [1.243 to 2.263]
Statistical Analysis 15: Comparison: Genotype 3; The statistical analysis is presented for weight per 10 kg. The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 1.384, 95% CI 2-sided [1.166 to 1.641]
Statistical Analysis 16: Comparison: Genotype 3; The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.090, 95% CI 2-sided [1.421 to 3.074]
Statistical Analysis 17: Comparison: Genotype 3; The statistical analysis is presented for liver fibrosis (no cirrhosis vs cirrhosis). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0006, Regression, Logistic; Odds Ratio (OR) = 0.288, 95% CI 2-sided [0.141 to 0.588]
Statistical Analysis 18: Comparison: Genotype 3; The statistical analysis is presented for liver fibrosis (not assessed/missing vs cirrhosis). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0013, Regression, Logistic; Odds Ratio (OR) = 0.247, 95% CI 2-sided [0.106 to 0.579]
Statistical Analysis 19: Comparison: Genotype 3; [analysis description as in outcome 19, analysis 8]; Test type: Superiority or Other; p = 0.0062, Regression, Logistic; Odds Ratio (OR) = 0.959, 95% CI 2-sided [0.931 to 0.988]
Statistical Analysis 20: Comparison: Genotype 3; The statistical analysis is presented for cumulative ribavirin dose per 10000 mg, first 12 weeks. The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including cumulative dose of peginterferon and ribavirin up to Week 12), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 0.708, 95% CI 2-sided [0.568 to 0.881]
Statistical Analysis 21: Comparison: Genotype 1; The statistical analysis is presented for age per 10 years. The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.434, 95% CI 2-sided [1.288 to 1.596]
Statistical Analysis 22: Comparison: Genotype 1; The statistical analysis is presented for HCV RNA at BL in log10 (IU/mL). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.475, 95% CI 2-sided [1.260 to 1.726]
Statistical Analysis 23: Comparison: Genotype 1; The statistical analysis is presented for treatment duration after VR in weeks. The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.963, 95% CI 2-sided [0.956 to 0.970]
Statistical Analysis 24: Comparison: Genotype 1; The statistical analysis is presented for cumulative PEG-IFN alfa-2a dose per 1000 ug. The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.195, 95% CI 2-sided [1.120 to 1.275]
Statistical Analysis 25: Comparison: Genotype 2; [analysis description as in outcome 19, analysis 21]; Test type: Superiority or Other; p = 0.0316, Regression, Logistic; Odds Ratio (OR) = 1.567, 95% CI 2-sided [1.040 to 2.359]
Statistical Analysis 26: Comparison: Genotype 2; The statistical analysis is presented for sex (male vs female). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0024, Regression, Logistic; Odds Ratio (OR) = 4.495, 95% CI 2-sided [1.701 to 11.879]
Statistical Analysis 27: Comparison: Genotype 2; The statistical analysis is presented for BMI in kg/m^2. The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0247, Regression, Logistic; Odds Ratio (OR) = 1.112, 95% CI 2-sided [1.014 to 1.219]
Statistical Analysis 28: Comparison: Genotype 2; [analysis description as in outcome 19, analysis 22]; Test type: Superiority or Other; p = 0.0258, Regression, Logistic; Odds Ratio (OR) = 1.844, 95% CI 2-sided [1.077 to 3.158]
Statistical Analysis 29: Comparison: Genotype 3; [analysis description as in outcome 19, analysis 21]; Test type: Superiority or Other; p = 0.0009, Regression, Logistic; Odds Ratio (OR) = 1.660, 95% CI 2-sided [1.232 to 2.235]
Statistical Analysis 30: Comparison: Genotype 3; The statistical analysis is presented for weight per 10 kg. The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0045, Regression, Logistic; Odds Ratio (OR) = 1.255, 95% CI 2-sided [1.073 to 1.467]
Statistical Analysis 31: Comparison: Genotype 3; [analysis description as in outcome 19, analysis 22]; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 2.086, 95% CI 2-sided [1.434 to 3.034]
Statistical Analysis 32: Comparison: Genotype 3; The statistical analysis is presented for liver fibrosis (no cirrhosis vs cirrhosis). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0010, Regression, Logistic; Odds Ratio (OR) = 0.318, 95% CI 2-sided [0.160 to 0.630]
Statistical Analysis 33: Comparison: Genotype 3; The statistical analysis is presented for liver fibrosis (not assessed/missing vs cirrhosis). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between treatment exposure and baseline factors available in at least 90% of participants (including total cumulative dose of peginterferon and ribavirin), in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0021, Regression, Logistic; Odds Ratio (OR) = 0.275, 95% CI 2-sided [0.121 to 0.626]
Statistical Analysis 34: Comparison: Genotype 3; [analysis description as in outcome 19, analysis 23]; Test type: Superiority or Other; p = 0.0064, Regression, Logistic; Odds Ratio (OR) = 0.962, 95% CI 2-sided [0.935 to 0.989]
Statistical Analysis 35: Comparison: Genotype 1; The statistical analysis is presented for age per 10 years. The logistic regression analysis for relapse 24 weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1.391, 95% CI 2-sided [1.245 to 1.553]
Statistical Analysis 36: Comparison: Genotype 1; The statistical analysis is presented for HCV RNA at BL in log10(IU/mL). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0029, Regression, Logistic; Odds Ratio (OR) = 1.295, 95% CI 2-sided [1.092 to 1.535]
Statistical Analysis 37: Comparison: Genotype 1; The statistical analysis is presented for On-treatment response (RVR vs no RVR/EVR). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.109, 95% CI 2-sided [0.050 to 0.236]
Statistical Analysis 38: Comparison: Genotype 1; The statistical analysis is presented for on-treatment response (cEVR vs no RVR/EVR). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0014, Regression, Logistic; Odds Ratio (OR) = 0.320, 95% CI 2-sided [0.159 to 0.645]
Statistical Analysis 39: Comparison: Genotype 1; The statistical analysis is presented for on-treatment response (pEVR vs no RVR/EVR). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.5390, Regression, Logistic; Odds Ratio (OR) = 1.248, 95% CI 2-sided [0.616 to 2.528]
Statistical Analysis 40: Comparison: Genotype 2; [analysis description as in outcome 19, analysis 35]; Test type: Superiority or Other; p = 0.0223, Regression, Logistic; Odds Ratio (OR) = 1.604, 95% CI 2-sided [1.069 to 2.405]
Statistical Analysis 41: Comparison: Genotype 2; The statistical analysis is presented for sex (male vs female). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0056, Regression, Logistic; Odds Ratio (OR) = 4.444, 95% CI 2-sided [1.547 to 12.766]
Statistical Analysis 42: Comparison: Genotype 2; The statistical analysis is presented for weight per 10 kg. The logistic regression analysis for relapse 24 weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0267, Regression, Logistic; Odds Ratio (OR) = 1.403, 95% CI 2-sided [1.040 to 1.892]
Statistical Analysis 43: Comparison: Genotype 2; The statistical analysis is presented for on-treatment response, combined (RVR vs no RVR). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0018, Regression, Logistic; Odds Ratio (OR) = 0.226, 95% CI 2-sided [0.089 to 0.575]
Statistical Analysis 44: Comparison: Genotype 3; [analysis description as in outcome 19, analysis 35]; Test type: Superiority or Other; p = 0.0083, Regression, Logistic; Odds Ratio (OR) = 1.529, 95% CI 2-sided [1.116 to 2.097]
Statistical Analysis 45: Comparison: Genotype 3; [analysis description as in outcome 19, analysis 42]; Test type: Superiority or Other; p = 0.0028, Regression, Logistic; Odds Ratio (OR) = 1.285, 95% CI 2-sided [1.090 to 1.515]
Statistical Analysis 46: Comparison: Genotype 3; [analysis description as in outcome 19, analysis 36]; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 2.061, 95% CI 2-sided [1.401 to 3.032]
Statistical Analysis 47: Comparison: Genotype 3; The statistical analysis is presented for liver fibrosis (no cirrhosis vs cirrhosis). The logistic regression analysis for relapse 24 Weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0019, Regression, Logistic; Odds Ratio (OR) = 0.327, 95% CI 2-sided [0.162 to 0.662]
Statistical Analysis 48: Comparison: Genotype 3; The statistical analysis is presented for liver fibrosis (not assessed/missed vs cirrhosis). The logistic regression analysis for relapse 24 weeks after EOT was performed for association between on-treatment response and baseline factors available in at least 90% of participants, in naive HCV mono-infected mTRT participants receiving PEG-IFN alfa-2a; Test type: Superiority or Other; p = 0.0086, Regression, Logistic; Odds Ratio (OR) = 0.320, 95% CI 2-sided [0.137 to 0.749]
Statistical Analysis 49: Comparison: Genotype 3; [analysis description as in outcome 19, analysis 43]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 0.247, 95% CI 2-sided [0.138 to 0.441]

20. Secondary Outcome: Percentage of Participants With Relapse After Modified End of Treatment Response by Genotype in Per Protocol Population at 24 Weeks After End of Treatment
Description: Participants whose last test result in the follow-up time window showed mVR were considered to have maintained their mEOT-R. Participants whose last test result in the respective follow-up time window did not show mVR, or who did not have a test result in the respective follow-up time window but whose last follow-up test result before the time window did not show mVR, were considered to have relapsed. Only participants with mEOT-R who had a HCV RNA measurement in the follow-up time window (without use of backward imputation), or whose last HCV RNA measurement at a follow-up time point before the time window did not show mVR, were included in the calculations. The percentage of participants with relapse is reported in treatment naive PP population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number; unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 1530 | 195 | 445 | 89 | 10 | 3
Percentage of participants | 26.6 | 10.8 | 16.6 | 24.7 | 0.0 | 0.0

21. Secondary Outcome: Percentage of Participants With Predictive Values of Virological Response by Week 2 on Modified Sustained Virological Response by Genotype After Treatment Initiation in Modified All-Treated Population
Description: The probability that a participant who developed VR by Wk 2 also achieved mSVR at 24 weeks after EOT was called the PPV of the VR by Wk 2 for mSVR. The probability that a participant who failed to develop VR by Wk 2 and also failed to achieve mSVR at 24 weeks after EOT was called the NPV of the VR by Wk 2 for mSVR. Predictive Values of VR was reported in treatment naive HCV mono-infected mTRT population receiving PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 1590 | 152 | 335 | 82 | 6 | 3
Percentage of participants
  At Week 2, PPV | 65.7 [57.3 to 73.5] | 89.7 [79.9 to 95.8] | 71.3 [61.8 to 79.6] | 73.3 [44.9 to 92.2] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0]
  At Week 2, NPV | 61.0 [58.5 to 63.5] | 35.7 [25.6 to 46.9] | 47.6 [40.9 to 54.3] | 65.7 [53.1 to 76.8] | 25.0 [0.6 to 80.6] | 50.0 [1.3 to 98.7]

22. Secondary Outcome: Percentage of Participants With Predictive Values of Virological Response by Week 2 on Modified Sustained Virological Response by Genotype After Treatment Initiation in Per-Protocol Population
Description: The probability that a participant who developed VR by Wk 2 and also achieved mSVR at 24 weeks after EOT was called the PPV of the VR by Wk 2 for mSVR. The probability that a participant who failed to develop VR by Wk 2 and also failed to achieve mSVR at 24 weeks after EOT was called the NPV of the VR by Wk 2 for mSVR. Predictive values of VR are reported in treatment naive HCV mono-infected PP population who received PEG-IFN alfa-2a. The EOT was 12, 24, 48 or 72 weeks after initiation of treatment.
Time Frame: At 24 weeks after EOT
Population: The PP population included all participants who met the inclusion/exclusion criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Number analyzed (Participants) | 1327 | 131 | 298 | 70 | 5 | 1
Percentage of participants
  At Week 2, PPV | 68.3 [59.3 to 76.4] | 91.8 [81.9 to 97.3] | 72.0 [62.1 to 80.5] | 69.2 [38.6 to 90.9] | 50.0 [1.3 to 98.7] | 100.0 [2.5 to 100.0]
  At Week 2, NPV | 60.0 [57.2 to 62.8] | 32.9 [22.1 to 45.1] | 46.0 [38.9 to 53.2] | 63.2 [49.3 to 75.6] | 0.0 [0.0 to 70.8] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: Up to 24 Weeks after EOT. The EOT is 12, 24, 48 or 72 weeks after initiation of treatment.
Description: Documentation of adverse event/serious adverse event was not within scope of this study. Serious Adverse Drug Reactions (SADRs) were to be reported spontaneously through spontaneous reporting system for marketed drugs. In most SADRs, the study number was missing on form; thus it could not be assigned to study and no data was available for reporting
Arm/Group | Genotype 1 | Genotype 2 | Genotype 3 | Genotype 4 | Genotype 5/6 | Genotype Unknown
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.